CLINICAL TRIAL: NCT05033561
Title: A Phase III Open-label Randomized Controlled Study to Evaluate the Safety and Immunogenicity of nOPV2 at Different Intervals of Administration in Infants
Brief Title: Study to Evaluate Safety and Immunogenicity of nOPV2 at Different Intervals in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: nOPV2-002-ABMG
Record Dates: First submitted 2021-08-19; First posted 2021-09-05 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-04

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2 doses, 1 week apart (Experimental): Administration of 2 doses of nOPV2, 1 week apart
  Interventions: Biological: nOPV2
- 2 doses, 2 week apart (Experimental): Administration of 2 doses of nOPV2, 2 weeks apart
  Interventions: Biological: nOPV2
- 2 doses, 4 week apart (Active Comparator): Administration of 2 doses of nOPV2, 4 weeks apart
  Interventions: Biological: nOPV2

INTERVENTIONS:
Biological: nOPV2 — Novel Oral Poliomyelitis Type 2 Vaccine

SUMMARY:
Study to determine immunogenicity and safety following administration of 2 doses of novel oral poliovirus vaccine type 2 (nOPV2) given at different intervals of 1 week or 2 weeks or the standard 4-week interval in infants

DETAILED DESCRIPTION:
This will be a multicenter, randomized, controlled, open-label, parallel-group Phase III study in healthy infants aged 6 to 8 weeks who have never been vaccinated against poliomyelitis. Approximately 900 infants will be included in the study and randomized with a 1:1:1 ratio to the following treatment groups:

* Group A: approximately 300 subjects to receive 2 doses of nOPV2 administered 1 week apart, at Day 0 and Day 7;
* Group B: approximately 300 subjects to receive 2 doses of nOPV2 administered 2 weeks apart, at Day 0 and Day 14;
* Group C (control group): approximately 300 subjects to receive 2 doses of nOPV2 administered 4 weeks apart, at Day 0 and Day 28. A total of 4 on-site visits are planned. Approximately 7 days after each administration of study vaccine, a phone call or on-site visit will be performed to monitor subjects' safety and review with the subject's parent(s)/guardian(s) any solicited AEs reported in the electronic diary card. All subjects will have a safety follow-up phone call 6 months after the last dose of study vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 6 to 8 weeks with birth weight > 2,500 g.
2. Healthy infants without obvious medical conditions like immunodeficiency diseases, severe congenital malformations, severe neurological diseases or any other disease that require high doses of corticosteroids or immunotherapies that preclude the subject from participating in the study as established by the medical history and physical examination.
3. Written informed consent obtained from 1 or 2 parent(s) or legal guardian(s) as per country regulations.

Exclusion Criteria:

1. Infants who have received previous vaccination against poliomyelitis.
2. Infants with anyone under 5 years of age in their household (living in the same house or apartment unit) who does not have the complete "age appropriate" vaccination status with respect to poliovirus vaccines at the time of study vaccine administration according to the Dominican Republic National Immunization Program (NIP).
3. Infants having a member of their household (living in the same house or apartment unit) who is under 6 months of age at the moment of study vaccine administration.
4. Infants having a member of their household (living in the same house or apartment unit) who has received oral poliomyelitis vaccine (OPV) in the previous 3 months before study vaccine administration.
5. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus infection in the potential participant or any member of the subject's household.
6. Family history of congenital or hereditary immunodeficiency.
7. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
8. Known allergy to any component of the study vaccine or to any antibiotics that share molecular composition with the nOPV2 vaccine.
9. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
10. Acute severe febrile illness on the day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all inclusion criteria are met.).
11. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.
12. Infants from multiple births or born prematurely (< 37 weeks of gestation)

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 905 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Dominican Republic (2):
  - Clinica Cruz Jiminián, Santo Domingo
  - Hospital Universitario Maternidad Nuestra Señora de la Altagracia, Santo Domingo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivera Mejia L, Pena Mendez L, Bandyopadhyay AS, Gast C, Mazara S, Rodriguez K, Rosario N, Zhang Y, Mainou BA, Jimeno J, Aguirre G, Ruttimann R. Safety and immunogenicity of shorter interval schedules of the novel oral poliovirus vaccine type 2 in infants: a phase 3, randomised, controlled, non-inferiority study in the Dominican Republic. Lancet Infect Dis. 2024 Mar;24(3):275-284. doi: 10.1016/S1473-3099(23)00519-4. Epub 2023 Dec 15. PMID 38109921

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Administration of 2 doses of nOPV2, 1 week apart
  nOPV2: Novel Oral Poliomyelitis Type 2 Vaccine
- Group B: Administration of 2 doses of nOPV2, 2 weeks apart
  nOPV2: Novel Oral Poliomyelitis Type 2 Vaccine
- Group C: Administration of 2 doses of nOPV2, 4 weeks apart
  nOPV2: Novel Oral Poliomyelitis Type 2 Vaccine
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 302 | 300 | 303
Completed | 297 | 297 | 298
Not Completed | 5 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Group A: Administration of 2 doses of nOPV2, 1 week apart
- Group B: Administration of 2 doses of nOPV2, 2 weeks apart
- Group C: Administration of 2 doses of nOPV2, 4 weeks apart
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 302 | 300 | 303 | 905
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 302 | 300 | 303 | 905
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 138 | 146 | 418
  Male | 168 | 162 | 157 | 487
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 1 | 1 | 3
  Mixed Race | 301 | 299 | 301 | 901
  Black or African American | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Dominican Republic | 302 | 300 | 303 | 905

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate at 1, 2 & 4 Weeks Interval
Description: Cumulative seroconversion rate of type 2 polio neutralizing antibodies 28 days following administration of 2 doses of nOPV2 in 1-week, 2-week and 4-weeks interval to infants 6 to 8 weeks of age
Time Frame: Up to max 8 weeks
Population: Per Protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 291 | 294 | 295
Participants | 253 | 269 | 277
Statistical Analysis 1: Comparison: Group A vs Group C; This study was designed to demonstrate the non-inferiority of Group A (1-week interval nOPV2 administration) and Group B (2-weeks interval nOPV2 administration) versus Group C (standard 4-week interval); Test type: Non-Inferiority — Non-inferiority would be verified if the lower bound of the two-sided 95% CI around each difference (shorter interval minus standard interval) is greater than -10%; p = 0.05, Miettinen-Nurminen — This is the nominal alpha level for the two-sided confidence interval comparison; Pairwise comparisons with two-sided Miettinen-Nurminen confidence intervals
Statistical Analysis 2: Comparison: Group B vs Group C; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Miettinen-Nurminen — This is the nominal alpha level for the two-sided confidence interval comparison; Pairwise comparisons with two-sided Miettinen-Nurminen confidence intervals

2. Secondary Outcome: Neutralizing Antibodies at 1, 2 & 4 Week Interval
Description: Geometric mean titers of type 2 polio neutralizing antibodies at Day 0 and 28 days after the second dose of nOPV2 when administered 1, 2 & 4 weeks apart.
Time Frame: Up to max 8 weeks
Population: Per Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 291 | 294 | 295
titers
  Day 0 | 10.7 [8.5 to 13.5] | 11.5 [9 to 14.7] | 10.2 [8.1 to 12.9]
  28 days after 2nd dose | 1232.3 [909 to 1670.5] | 1726.3 [1252.1 to 2380.1] | 2327.6 [1654.3 to 3275.2]
Statistical Analysis 1: Comparison: Group A vs Group C; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Miettinen-Nurminen — This is the nominal alpha level for the two-sided confidence interval comparison; Pairwise comparisons with two-sided Miettinen-Nurminen confidence intervals
Statistical Analysis 2: Comparison: Group B vs Group C; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Miettinen-Nurminen — This is the nominal alpha level for the two-sided confidence interval comparison; Pairwise comparisons with two-sided Miettinen-Nurminen confidence intervals

3. Secondary Outcome: Serious Adverse Events (SAEs) and Important Medical Events (IMEs)
Description: Number of participants experiencing SAEs and IMEs from the date of informed consent throughout the study period in all groups by severity and by causal association.
Time Frame: 6 months
Population: Total Vaccinated Population. Please note that for the safety analysis, subjects were classified according to the actual administration interval received per the Statistical Analysis Plan. Thus, 4 patients randomized into Group A were assigned to Group B for safety analysis tables.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 298 | 304 | 303
Participants
  Death | 0 | 0 | 1
  Hospitalization | 8 | 7 | 9
  Birth defect | 1 | 1 | 0

4. Secondary Outcome: Solicited Adverse Events (AEs)
Description: Number of participants experiencing mild, moderate and severe solicited AEs (fever, vomiting, abnormal crying, drowsiness, loss of appetite, diarrhea and irritability) for 7 days after each dose of study vaccine in all groups.
Time Frame: Up to max 5 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 294 | 304 | 303
Participants
  Abnormal crying | 84 | 90 | 83
  Diarrhea | 44 | 50 | 40
  Drowsiness | 25 | 38 | 36
  Fever | 134 | 147 | 139
  Irritability | 31 | 45 | 41
  Loss of Apetite | 36 | 49 | 38
  Vomiting | 45 | 75 | 62

5. Secondary Outcome: Unsolicited Adverse Events (AEs)
Description: Number of participants experiencing mild, moderate, and severe solicited AEs (fever, vomiting, abnormal crying, drowsiness, loss of appetite, diarrhea, and irritability) for 28 days after each dose of study vaccine in all groups.
Time Frame: Up to max 8 weeks
Population: Total Vaccinated Population. Please note that for the safety analysis, subjects were classified according to the actual administration interval received per the Statistical Analysis Plan (SAP). Thus, 4 patients randomized into Group A were assigned to Group B for safety analysis tables.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 298 | 304 | 303
Participants
  Respiratory disorders | 13 | 10 | 11
  Infections | 9 | 10 | 14
  Gastrointestinal disorders | 3 | 13 | 9
  Musculoskeletal and connective tissue disorders | 0 | 0 | 3
  Skin disorders | 0 | 2 | 1
  Congenital disorders | 0 | 1 | 1
  Nervous system disorders | 0 | 1 | 0
  General disorders | 1 | 8 | 6

ADVERSE EVENTS:
Time Frame: 6 months
Description: Assessments were performed on the Total Vaccinated Population (TVP). Please note that for the safety analysis, subjects were classified according to the actual administration interval received per the Statistical Analysis Plan. Thus, 4 patients randomized into Group A were assigned to Group B for safety analysis tables.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/304 | 1/303
Serious Adverse Events (participants affected / at risk) | 8/298 | 7/304 | 9/303
Other Adverse Events (participants affected / at risk) | 217/298 | 247/304 | 238/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=298) | Group B (N=304) | Group C (N=303)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 5 (5)
Bronchiolitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hereditary haemolytic anemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hereditary spherocytosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=298) | Group B (N=304) | Group C (N=303)
Abnormal crying (General disorders) | 84 (102) | 92 (144) | 83 (123)
Diarrhoea (Gastrointestinal disorders) | 46 (59) | 56 (80) | 44 (64)
Drowsiness (Nervous system disorders) | 25 (28) | 38 (47) | 36 (49)
Fever (General disorders) | 135 (153) | 152 (182) | 144 (164)
Irritability (Nervous system disorders) | 31 (41) | 46 (65) | 41 (55)
Loss of apetite (Gastrointestinal disorders) | 36 (42) | 49 (53) | 38 (45)
Vomiting (Gastrointestinal disorders) | 45 (65) | 81 (118) | 65 (97)
Nasal congestion (Infections and infestations) | 11 (11) | 2 (2) | 4 (4)
Rhinorrhoea (Infections and infestations) | 2 (2) | 5 (5) | 6 (6)
Cough (Infections and infestations) | 2 (2) | 5 (5) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Amoebic Dysentery (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI and/or the Institution are not entitled to publish or present any study information, either partial or complete, without written approval by FIDEC.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT05033561/Prot_SAP_000.pdf